CLINICAL TRIAL: NCT06133231
Title: A Feasibility and Acceptability Study (FAST) to Optimize Research Methodology in a Multinutrient Study of Racially and Ethnically Diverse Children With ADHD and Emotional Dysregulation
Brief Title: Optimizing Research With Diverse Families - Feasibility and Acceptability Study (FAST)
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeanette Johnstone, Associate Professor, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00024336
Record Dates: First submitted 2023-06-12; First posted 2023-11-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Emotional Dysfunction; Irritable Mood
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Minerals; Amino Acids; Antioxidants

STUDY DESIGN:
Intervention Model Description: Feasibility of using multinutrient intervention with previously under-represented populations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multinutrient (Experimental): All participants will take the active multinutrient treatment
  Interventions: Dietary Supplement: Multinutrients; a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants

INTERVENTIONS:
Dietary Supplement: Multinutrients; a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants — Participants will take 2-4 capsules of EMP+ Advanced per day (max 8 capsules) for eight weeks.
  Other Names: EmpowerPlus (EMP+) Advanced

SUMMARY:
Evaluate feasibility and acceptability of recruiting Black and Hispanic families for an open label clinical trial of multinutrients while collecting real-time parent-reported child behavior data and collecting at-home biospecimens to explore their potential as biomarkers, in a study of pediatric ADHD.

DETAILED DESCRIPTION:
This study will test the feasibility of recruiting and completing a multinutrient trial with racially and ethnically diverse participants (N=30), focused on Black and Hispanic families, and the acceptability of the intervention, and refined collection methods. The 8-week, open-label, study will evaluate the feasibility and acceptability of collecting (a) real-time ecological momentary assessment (EMA) data on child's target behavior problem, as identified by parent and (b) two types of bio-specimens (blood and urine) collected at home while taking the multinutrients daily.

ELIGIBILITY:
Inclusion Criteria:

* Children, ages 6-17 years at enrollment, with suspected or definite ADHD based on parent report in a majority of families that identify as Black or Hispanic or multicultural
* Meet criteria on Child and Adolescent Symptom Inventory-5 (CASI-5) ADHD scale (6+ symptoms ≥ 2), occurring in >1 setting, plus one impairing irritability symptom (≥2) from Oppositional Defiant Disorder (ODD) or Disruptive Mood Dysregulation Disorder (DMDD) subscale
* Able and willing to swallow up to 8 pills per day
* Medication free for 2 weeks prior to baseline
* Willing to use Tasso® OnDemand SST+ to collect blood at home and filter cards to provide urine samples
* Able to communicate in English
* Parent/care giver identifies child as Black/African American or Hispanic/Latina/o or more than one race (target 70-100%)

Exclusion Criteria:

* Neurological disorders
* Medical conditions (e.g. cancer, kidney or liver disease, diabetes, hyperthyroidism)
* Psychiatric conditions requiring hospitalization
* Allergy to any supplement ingredient
* In people with a uterus: sexually active, pregnancy or suspected pregnancy
* Abnormality of mineral metabolism

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility measured by count of consumed multinutrients | Week 4, Week 8
  Feasibility will be determined based on consumption of the number of capsules determined to be beneficial based on parent and child report of symptom improvement or side effects, typically 2-4 capsules per day (up to max of 8) and achieved when greater than or equal to 75% of recommended doses have been consumed as measured at week 4 and at week 8 by pill count.
Abbreviated Acceptability Rating Profile - 7 questions on a 6-point Likert scale | Week 8
  Acceptability of taking the multinutrients will be measured through 7 questions with a 6-point Likert scale (range: Strongly Disagree to Strongly Agree). Acceptability will be achieved if greater than or equal to 70% of children and parents report that taking the capsuled multinutrients is acceptable, at or above the "Agree" range - scores of 5 or 6.

SECONDARY OUTCOMES:
Feasibility of Capillary Blood Collection | Baseline
  Feasibility will be measured as the frequency/percentage of children who provide capillary blood sample using the self-administered Tasso® OnDemand SST+ device. Device use will be considered feasible if greater than or equal to 70% of children provide the sample.
Acceptability of Capillary Blood Collection | Baseline
  Child acceptability will be a 10-point Visual Analog Scale (VAS) and brief quantitative feedback regarding the blood collection process for children. Parent acceptability will be measured using a 6-point Likert scale with 4 items. Acceptability will be achieved if greater than or equal to 70% of children respond with scores of 1 to 5 ("It was okay, fine" and "It was good, no problem") and 70% of parents report that using the Tasso device is acceptable at or above the "Agree" range - scores of 5 or 6.
Feasibility of Collecting 24-hour Urine | 4x on one day only to reflect 24-hour urine collection - Baseline, Week 8
  Feasibility will be measured as the frequency/percentage who provide at least 3 of the 4 urine samples in the 24-hour period, measured at two time points: baseline and week 8. At-home collection of dried urine samples will be considered feasible if greater than or equal to 70% of children provide the sample.
Acceptability of Collecting 24-hour Urine | Week 8
  Child acceptability will be a 6-point Likert scale of 4 questions with a visual analog scale and brief qualitative feedback regarding the urine collection process (range: Strongly Disagree to Strongly Agree). Parent acceptability will be a 6-point Likert scale with 4 questions (range: Strongly Disagree to Strongly Agree). Acceptability will be achieved if greater than or equal to 70% of children and parents report that the at-home dried urine collection method is acceptable at or above the "Agree" range - scores of 5 or 6.
Child and Adolescent Symptom Inventory (CASI-5) | Baseline, Week 4, Week 8
  The CASI-5 is based on the DSM-5 symptom criteria. The subscales of ADHD, Oppositional Defiant Disorder (ODD), Disruptive Mood Dysregulation Disorder (DMDD) and peer conflict will be combined into a total composite score; range is 0-3 (never, sometimes, often, very often). Higher scores represent a worse outcome. These scores will be used to look for signals of change over time.
Clinical Global Impression - Improvement (CGI-I) | Week 4, Week 8
  The clinician-rated CGI-Improvement (CGI-I) is a subscale of the CGI that rates overall improvement of symptoms based on all relevant data. Item range is 1-7 (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse); lower score is better. A treatment responder is defined as a participant who is rated a 1 or 2 on the CGI-I. These scores will be used to look for signals of change over time.
Clinical Global Impression - Severity (CGI-S) | Baseline, Week 8
  The CGI-Severity (CGI-S) subscale scores compared at the two time points. Item range is 1-7 (normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among the most extremely ill patients); lower score is better; most participants will be a 4 or 5 at baseline. These scores will be used to look for signals of change over time.
Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA-24) | Baseline and Week 8
  Parent report of child's 24-hour dietary intake The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool is a free, web-based tool. ASA-24 enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records. Parent will report of child's 24-hour dietary intake at baseline and at week 8. These scores will be used to look control for dietary differences at baseline and to control for dietary changes over time.
Parent Target Problem (PTP) using Ecological Momentary Assessment (EMA) | Baseline to Week 8, daily
  Parents are prompted to nominate the child's most impairing behavior and qualitatively describe it, then quantitatively report: 1) frequency: how often the problem behavior occurs (times a day, week), 2) duration: how long the problem behavior lasts when it occurs, 3) intensity: how impairing is it on a scale of 1 to 10. Reporting on the behavior will occur every day, at home, in response to a pre-populated questionnaire designed to be completed in one-two minutes or less, which may be accessed on a mobile phone, tablet or computer. Data will be collected for 60 days. Data will be used to detect signals of change over time.
Feasibility of Collecting Real-Time EMA Parent Target Problem (PTP) | Week 4, Week 8
  Feasibility will explore the average number of timepoints the parent/caregiver provided EMA data during the prior weeks before their week 4 and week 8 visit. At-home completion of parent-target-problems will be considered feasible if parents respond to greater than or equal to 70% of the prompts.
Acceptability of Collecting Real-Time EMA Parent Target Problem (PTP) | Week 8
  Acceptability will be a 6-point Likert scale with 3 questions and brief qualitative feedback regarding the EMA data collection process (range: Strongly Disagree to Strongly Agree). Acceptability will be achieved if greater than or equal to 70% of parents report that the EMA data collection method is acceptable at or above the "Agree" range, scores of 5 or 6.
Pediatric Adverse Events Rating Scale (PAERS) | Baseline, Week 4, Week 8
  Parent will report on possible side effects using PAERS to respond to presence, frequency and severity of 43-items, including: headache, dry mouth, sleep disruptions, nausea, irritability, fatigue, anxiety, changes in appetite, skin rash, migraines, and other (parents specify the symptom). Occurrence of these data will be reported at week 4 and 8.
Reasons for Dropout | Before week 7
  In order to assess for acceptability, parents whose children drop out of the study before week 7 will be contacted to ask, qualitatively, their reason for dropout. The responses will be recorded and reported .

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Johnstone, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States